CLINICAL TRIAL: NCT07056595
Title: Finerenone in Patients With IgA-nephropathy: Prospective Interventional Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Botkin Hospital (Other)
Responsible Party: Principal Investigator, Evgeny Shutov, Senior Researcher, Botkin Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEC-6/13052025
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: IgA Nephropathy (IgAN)
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — finerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iRAS (Experimental)
  Interventions: Drug: Finerenone
- iSGLT2 (Experimental)
  Interventions: Drug: Finerenone
- iRAS+iSGLT2 (Experimental)
  Interventions: Drug: Finerenone

INTERVENTIONS:
Drug: Finerenone — Finerenone is a new nonsteroidal mineralocorticoid receptor antagonist. Planned dose - 10 mg/day

SUMMARY:
: IgA-nephropathy is the most common glomerulonephritis with the unfavorable prognosis in patients with persistent albuminuria. Finerenone is a new nonsteroidal mineralocorticoid receptor antagonist that has demonstrated efficacy in reducing albuminuria in patients with CKD and type 2 diabetes in two major trials, FIGARO-DKD and FIDELIO. This finding supported the approval of finerenone by the U.S. Food and Drug Administration (FDA) for the treatment of chronic kidney disease (CKD). A subgroup analysis in the pooled FIDELITY trial demonstrated that in patients with CKD stages 1-4 and type 2 diabetes (T2D), the cardio- and nephroprotective effects of finerenone were independent of concomitant therapy with SGLT-2 inhibitors or GLP-1 receptor agonists. Thus, the role of finerenone in slowing CKD progression in T2D can be considered well-established. Given its albuminuria-reducing effects, finerenone is being investigated in multiple trials, including studies on non-diabetic kidney disease and IgA nephropathy, though no published results are available yet. In this trial finerenone will be used as a nephroprotective agent above standard treatment in terms of assessing adverse events and potential efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years) with the primary IgAN diagnosed by kidney biopsy;
* Treatment with stable doses of iRAS or/and iSGLT2 inhibitors for at least 3 months prior inclusion into the trial;
* Blood pressure < 140/90 mm Hg
* 24-hour urinary albumin excretion > 300 mg

Exclusion Criteria:

* Kidney transplantation in medical history
* Chronic hepatic disease, including hepatitis, malignant tumor, active malignancy;
* Heart failure with ejection fraction <40%;
* Acute myocardial infarction and/or stroke less then 3 months before including in trial;
* Presence ANCA in serum
* Ongoing immunosuppressive treatment
* eGFR < 20 ml/min
* Pregnancy and breastfeeding
* Uncontrolled blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-05-21 (Estimated); Study Completion 2026-05-21 (Estimated)

PRIMARY OUTCOMES:
Median change in albuminuria from baseline | 6 months
  24-hour urinary albumin excretion

OTHER OUTCOMES:
Median change in eGFR from baseline | 6 months
  calculated based on creatinine level

CONTACTS AND LOCATIONS:
Locations (1):
- Botkin Hospital, Moscow, Russia